CLINICAL TRIAL: NCT03369275
Title: Cellular Immunotherapy for Septic Shock (CISS2) A Phase II Randomized Controlled Trial
Brief Title: Cellular Immunotherapy for Septic Shock
Acronym: CISS2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Institute for Regenerative Medicine (OIRM) (Unknown); Stem Cell Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201706
Record Dates: First submitted 2017-08-28; First posted 2017-12-11 (Actual); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Septic Shock; Sepsis; Pathologic Processes; Shock; Infection; Systemic Inflammatory Response Syndrome; Inflammation
Keywords: Mesenchymal Stem Cells; Mesenchymal Stromal Cells; Randomized Controlled Trial; Cryopreserved; Allogeneic; Phase II
MeSH Terms: conditions — Shock, Septic; Sepsis; Pathologic Processes; Shock; Infections; Systemic Inflammatory Response Syndrome; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stromal Cells (MSCs) (Experimental): Intravenous infusion of 300 million Allogeneic, Bone Marrow-Derived Human Mesenchymal Stromal Cells
  Interventions: Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells
- Placebo (Placebo Comparator): Intravenous infusion of Placebo, with excipients
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells — Cryopreserved Allogeneic Bone Marrow-Derived Human Mesenchymal Stem Cells will be administered intravenously.
  Arms: Mesenchymal Stromal Cells (MSCs)
Other: Placebo — Placebo, with excipients, will be administered intravenously.
  Arms: Placebo

SUMMARY:
Septic shock is associated with substantial burden in terms of both mortality and morbidity for survivors of this illness. Pre-clinical sepsis studies suggest that mesenchymal stem (stromal) cells may modulate inflammation, enhance pathogen clearance and tissue repair and reduce death. Our team has completed a Phase I dose escalation and safety clinical trial that evaluated mesenchymal stem cells (MSCs) in patients with septic shock. The Cellular Immunotherapy for Septic Shock (CISS) trial established that MSCs appear safe and that a randomized controlled trial (RCT) is feasible. Based on these data, the investigators have planned a phase II RCT (CISS2) at several Canadian academic centres which will evaluate safety, signals for clinical efficacy, and continue to examine potential mechanisms of action and biological effects of MSCs in septic shock.

DETAILED DESCRIPTION:
Septic shock is a devastating illness and the most severe form of infection seen in the intensive care unit (ICU). It is characterized by cardiovascular collapse, failure of organs and is common with severe repercussions including a mortality of 20-40%. Survivors suffer long-term impairment in function and reduced quality of life (QOL). Despite decades of research examining different immune therapies, none has proven successful and supportive care remains the mainstay of therapy, at a cost of approximately 4-billion dollars in Canada annually. MSCs represent a potentially novel treatment for sepsis because in animal models, MSCs have been shown to modulate the immune system, increase pathogen clearance, restore organ function, and reduce death.

The Phase II multi-centre Cellular Immunotherapy for Septic Shock RCT (CISS2) will continue to evaluate safety, assess if there are signals for clinical efficacy and determine mechanisms of action and biological effects of MSCs in septic shock. To answer these aims, CISS2 will randomize 114 patients who are admitted to the ICU with septic shock to 300 million cryopreserved, allogeneic, bone marrow derived MSCs or placebo across 10 Canadian centres over approximately 2 years.

ELIGIBILITY:
Inclusion Criteria:

A participant must meet all three inclusion criteria to be eligible:

1. Admission to an Intensive Care Unit AND
2. Cardiovascular failure that is present within the first 24 hours of admission to the ICU and is defined by the requirement for at least 15 mcg/min of norepinephrine or at least 200 mcg/min of phenylephrine or at least 0.03 U/min of vasopressin, or a combination of norepinephrine and phenylephrine that is equivalent to the total required doses (e.g. norepinephrine 8 meq/min and phenylephrine 100 mcg/min) for at least 4 consecutive hours. Participants must still require vasopressor(s) at the time of MSC infusion to be eligible. AND
3. At least 1 additional organ failure, or organ hypoperfusion, as defined by the modified Multiple Organ Dysfunction Score (MODS). Criteria for organ dysfunction or organ hypoperfusion must be met within the first 24 hours of ICU admission. These include:

   1. Respiratory failure: mechanically ventilated with a positive end expiratory pressure (PEEP) of at least 5 cm H20, and a partial pressure of oxygen/fractional inspired oxygen concentration (P/F ratio) less than or equal to 200 on 2 separate occasions.
   2. Hematological failure: platelet count of less than or equal to 100 X 109 /L that has decreased by at least 50 x 109/L.
   3. Acute renal failure: acute renal insufficiency with a creatinine of greater than 200 umol/L that has increased by at least 50 umol/L, or the requirement for continuous renal replacement therapy, or for participants with known chronic renal failure but not on dialysis, a 50% increase in their baseline creatinine concentration.
   4. Organ hypoperfusion: a lactate of at least 4 mmol/L

Acute organ failures that meet eligibility criteria cannot have been present for more than 48 hours prior to admission to the ICU.

Exclusion Criteria:

1. Another form of shock (cardiogenic, hypovolemic, obstructive) that is considered by the treating critical care staff physician as the dominant cause of shock.
2. History of known chronic pulmonary hypertension with a WHO functional class of III or IV
3. History of severe chronic pulmonary disease requiring home oxygen
4. History of chronic severe cardiac disease including congestive heart failure or valvular dysfunction with a New York Heart Association Functional Class of III or IV, or severe ischemic heart disease with a Canadian Cardiovascular Society angina class score of III or IV.
5. History of severe chronic liver disease (Child class C)
6. Malignancy in the previous year (excluding resolved non-melanoma skin cancer). Participants will be excluded from the CISS2 trial if they have received any surgery, chemotherapy, or radiation for a malignancy in the previous 12 months.
7. Chronic immune suppression (chronic steroid use or chemotherapy)
8. Pregnant or lactating
9. Enrolment in another interventional study
10. Treating physicians' impression is that the participant is moribund and that death is imminent within the subsequent 12 hours of meeting eligibility criteria
11. Family, participant, or physician not committed to aggressive care. Any limitation of care will exclude the patient from enrolment in the CISS2 trial (ex: no intubation, no use of vasopressor agent(s), no renal support therapy).
12. Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2018-03 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
The reduction in days on mechanical ventilation, or renal replacement therapy, or vasopressors. | Through to 28 days post-randomization
  The number of days free from each of these support measures.
Incidence of treatment-emergent adverse events (Safety and tolerability) | Through to 28 days post-randomization

SECONDARY OUTCOMES:
Biological endpoints as markers of vascular permeability | At baseline, 1, 2, 3 and 7 days post-randomization
  Marker of vascular permeability (ex: Ang1 and 2), acute renal injury (ex: Urine TIMP2-IGFBP7, IL-18), muscle weakness (ex: micro RNA (miRNA) growth Differentiation Factor-15 and miR-181a)), mechanisms related to pathogen clearance (ex: cathelicidin, LL-37), and pro and anti-inflammatory cytokines (ex: IL-6, IL-8, IL-10, IL-1B and IL1-RA) related to potential MSC biological effects
Mortality | Through to 12 months post-randomization
  All-cause mortality
Organ Failure Scores | Through to 90 days post-randomization
  Sequential Organ Failure Assessment (SOFA) Score
Organ Support Measures | Through to 90 days post-randomization
  Duration of mechanical ventilation and/or vasopressor agents and/or dialysis/renal replacement therapy
Length of ICU Stay (in days) | Number of elapsed days from admission until ICU discharge, up to one year
  Time in ICU
Length of Hospital Stay (in days) | Number of elapsed days from admission until hospital discharge, up to one year
  Time in Hospital
Hospital Re-Admissions | At 28 days, 3 and 12 months post-randomization
Patient Reported Outcomes-FIM | 7 days and 6 months post-ICU discharge
  Functional Independence Measure (FIM)
Patient Reported Outcomes-SF 36 | 7 days and 6 months post-ICU discharge
  SF-36 Score

CONTACTS AND LOCATIONS:
Overall Officials: Lauralyn McIntyre, MD, Principal Investigator — The Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: Undecided